CLINICAL TRIAL: NCT05371912
Title: Enhancement of Behavioral and Cognitive Outcomes in Autism Spectrum Disorder Via Neurostimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christiana Care Health Services (Other)
Collaborators: Dupont Applied Biosciences (Industry)
Responsible Party: Principal Investigator, Mitra Assadi, Medical Director, Christiana Care Health Services
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DDD 604994
Record Dates: First submitted 2022-05-01; First posted 2022-05-12 (Actual); Results first posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: The patients will be randomized at the time of recruitment to either receiving left or right IPL stimulation. A shamming technique will be applied to the opposite hemisphere. Both the patient and the neuropsychologist obtaining and interpreting the outcome measures will be blinded regarding the hemispheric side of rTMS intervention. Only the clinician delivering the rTMS treatment will have a knowledge about the treatment targeting.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The TMS coil will be placed on the scalp at a 90 degree angle and will be turned on to create the perception of delivering the stimulation to the brain.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- left IPL stimulation (Active Comparator): half of the subjects will receive TMS on the left inferior parietal lobule.
  Interventions: Device: Trans Cranial Magnetic Stimulation
- right IPL stimulation (Active Comparator): half of the subjects will receive TMS on the right inferior parietal lobule.
  Interventions: Device: Trans Cranial Magnetic Stimulation

INTERVENTIONS:
Device: Trans Cranial Magnetic Stimulation — Repetitive transcranial magnetic stimulation (rTMS) is a non-invasive neurostimulation technique that alters cortical excitability by repeated induction of electromagnetic activity. FDA approved for depression, rTMS is a promising tool in the field of neuropsychiatry with an excellent safety profile.

SUMMARY:
Autism spectrum disorder (ASD) encompasses a range of limitations in reciprocal social and communicative milestones, as well as restrictive and/or repetitive patterns of behavior which lead to significant functional challenges impacting individuals throughout their lifespan. There are major shortcomings in the existing pharmacological interventions; they are of limited efficacy, target a subset of problematic behaviors, and fail to improve social cognition. To overcome these limitations and improve outcomes, the investigators study the use of neurostimulation to mitigate the social and cognitive manifestations of ASD.

DETAILED DESCRIPTION:
Repetitive transcranial magnetic stimulation (rTMS) is a non-invasive neurostimulation technique that alters cortical excitability by repeated induction of electromagnetic activity. FDA approved for depression, rTMS is a promising tool in the field of neuropsychiatry with an excellent safety profile. A prevailing hypothesis in ASD proposes that mirror neuron dysfunction in the inferior parietal lobule (IPL) contributes to the core deficits. The left and right IPL regions support different social and cognitive functions and moreover, are differentially impacted in ASD. Therefore, it can be expected that enhancing function of the IPL may produce positive but hemispheric-dependent effects on social cognition. The investigators long-term goal in this pilot proposal is to understand whether stimulating IPL with rTMS improves social and cognitive outcomes in ASD.

This research, which builds upon our proof-of-concept testing of 4 patients, proposes 10 sessions of rTMS stimulation of the IPL. Participants will be randomized to receive active stimulation to either the left or right-IPL (with sham stimulation to the contralateral side) in a prospective, double-blind protocol during which neither the subject nor the neuropsychologist obtaining and interpreting the outcome measures will have awareness of the rTMS group. For targeting the IPL, which correlates with the Brodmann areas 40/7 on the cortex, the investigators use disposable mapping caps, and for the purpose of blinding, the investigators use a standard shamming technique. Outcome measures include neuropsychological testing administered at baseline, after completion of TMS regime, and three months later. Within this design, the investigators have three aims:

Aim 1: Assess the differential effects of rTMS of the left versus right IPL on linguistic abilities and executive function in ASD. Hypothesis: rTMS stimulation of the IPL leads to long term potentiation and hence enhances cognitive performance in a hemispheric dependent manner with left-IPL stimulation enhancing linguistic ability and right-IPL stimulation enhancing executive function. To measure the effects, the investigators will use the Delis-Kaplan Executive Function System Verbal Fluency task (D-KEFS) and two elements of the NIH toolbox: Flanker: a test to measure the inhibitory and attentional facets of Executive Functioning. Dimensional Change Card Sort (DCCS): a task designed to assess cognitive flexibility. The investigators expect improvement in the Flanker and DCCS scores with right IPL stimulation and D-KEFS score improvement with left IPL stimulation.

Aim 2: Determine the effects of unilateral rTMS of the IPL on social/behavioral deficits in children and young adults with ASD. Hypothesis: rTMS simulation of the mirror neuron system potentiates similar improvements in social cognition despite hemispheric laterality via separate but related mechanisms. To measure the outcomes of right v/s left unilateral IPL stimulation, the investigators will use two standard scales and compare the numerical values before and after the intervention. The Social Responsiveness Scale - 2nd Edition (SRS2) and the Repetitive Behavior Scale-Revised (RRBs) are validated parent/caregiver-rated scale of social/communication deficits and restricted/repetitive behaviors respectively.

ELIGIBILITY:
Inclusion criteria

* Fulfilling the Diagnostic and Statistical Manual for Mental Disorders 5th edition (DSM-V) criteria for ASD and confirmed by Gilliam Asperger Disorder Scale (GADS)
* The patient exhibiting adequate understanding and cooperation for the procedure

Exclusion criteria

* Patients with ASD exhibiting significant anxiety or contact avoidance, precluding them from cooperating with the procedure
* Children with a known diagnosis of seizures
* Presence of any metallic implants or devices in the head or neck area
* Pregnant women

Ages: 5 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2024-02-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Mitra Assadi, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from outpatient clinics and community referrals. Eligible participants were randomized 1:1 to left-IPL or right-IPL rTMS.
Pre-assignment Details: All patients met the diagnostic criteria for autism spectrum disorder. We excluded all patients with history of seizures or metallic devices in the hedonic area.
Period: Overall Study
Arm/Group | Left IPL Stimulation | Right IPL Stimulation
Started | 8 | 8
Completed | 5 | 6
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Left IPL Stimulation: 8 subjects received TMS on the left inferior parietal lobule(IPL). The average age was 13.3 years. Gender: The participants were all male Race: black, white and Asian
- Right IPL Stimulation: 8 subjects received TMS on the right inferior parietal lobule(IPL).
  The average age was 13.3 years. Gender: 7 male and 1 female Race: black, white and Asian
- Total: Total of all reporting groups
Arm/Group | Left IPL Stimulation | Right IPL Stimulation | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 7 | 13
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 8 | 7 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 5 | 5 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Social Awareness [Mean (Standard Deviation); unit: total raw score (0-195; higher = worse)] — Social Responsiveness Scale, Second Edition (SRS-2), Parent/Caregiver form; 65 items scored 0-3; total raw score range 0-195. Higher scores = greater social impairment. This study reports raw totals (not T-scores). Instrument: SRS-2. Population: 5 drop outs
  total raw score (0-195; higher = worse)
    number analyzed (Participants) | 5 | 6 | 11
    (all) | 68 (9.823) | 79.667 (14.624) | 74.364 (13.515)
reciprocal rigid patterns of behavior [Mean (Standard Deviation); unit: total raw score (0-129; higher = worse)] — Repetitive Behavior Scale-Revised (RBS-R); 43 items scored 0-3; total raw score range 0-129. Higher scores = more severe restricted/repetitive behaviors. We report total raw scores. Population: 5 drop outs
  total raw score (0-129; higher = worse)
    number analyzed (Participants) | 5 | 6 | 11
    (all) | 75.8 (11.212) | 86.667 (14.334) | 81.727 (13.609)
verbal fluency [Mean (Standard Deviation); unit: scaled score ( higher = better)] — Delis-Kaplan Executive Function System (D-KEFS) Verbal Fluency; scores converted to age-normed scaled scores (mean 10, Standard Deviation(SD) 3). Higher scores = better verbal fluency/executive function. We report the Total Correct scaled score per the manual. Population: 5 drop outs
  scaled score ( higher = better)
    number analyzed (Participants) | 5 | 6 | 11
    (all) | 5.8 (3.384) | 8.5 (7.778) | 6.571 (4.650)
Executive function [Mean (Standard Deviation); unit: standard score (higher =better)] — NIH Toolbox Flanker Inhibitory Control and Attention; Age-Adjusted Standard Scores (mean 100, SD 15) reported. Higher scores = better inhibitory control/attention. Population: 5 drop outs
  standard score (higher =better)
    number analyzed (Participants) | 5 | 6 | 11
    (all) | 66.8 (14.025) | 86 (22.996) | 77.273 (21.062)
Executive Function [Mean (Standard Deviation); unit: standard score ( higher=better)] — NIH Toolbox Dimensional Change Card Sort (DCCS); Age-Adjusted Standard Scores (mean 100, SD 15) reported. Higher scores = better cognitive flexibility. Population: 5 drop outs
  standard score ( higher=better)
    number analyzed (Participants) | 5 | 6 | 11
    (all) | 77.4 (23.416) | 76.8 (23.784) | 77.1 (22.253)

OUTCOME MEASURES:

1. Primary Outcome: The Effects of rTMS on Reciprocal Social Awareness
Description: Social Responsiveness Scale, Second Edition (SRS-2), Parent/Caregiver form; 65 items scored 0-3; total raw score range 0-195. Higher scores = greater social impairment. This study reports raw totals (not T-scores). Instrument: SRS-2
Time Frame: at baseline and 5 weeks of rTMS
Population: Subjects were randomized to receive right or left IPL stimulation.
Measure: Mean (Standard Deviation); unit: total raw score (higher=worse)
Arm/Group | Left IPL Stimulation | Right IPL Stimulation
Number analyzed (Participants) | 5 | 6
total raw score (higher=worse)
  Baseline | 68 (9.823) | 79.667 (14.624)
  Week 5 | 64.2 (5.310) | 74 (16.505)

2. Primary Outcome: The Effects of rTMS on Reciprocal Rigid Patterns of Behavior
Description: Repetitive Behavior Scale-Revised (RBS-R); 43 items scored 0-3; total raw score range 0-129. Higher scores = more severe restricted/repetitive behaviors. We report total raw scores.
Time Frame: at baseline and 5 weeks of rTMS
Population: Subjects were randomized to receive right or left IPL stimulation.
Measure: Mean (Standard Deviation); unit: total raw score (0-129; higher = worse)
Arm/Group | Left IPL Stimulation | Right IPL Stimulation
Number analyzed (Participants) | 5 | 6
total raw score (0-129; higher = worse)
  Baseline | 75.8 (11.212) | 86.667 (14.334)
  Week 5 | 75.4 (12.260) | 81.333 (12.879)

3. Secondary Outcome: The Effect of rTMS on Verbal Fluency
Description: Delis-Kaplan Executive Function System (D-KEFS) Verbal Fluency; scores converted to age-normed scaled scores (mean 10, SD 3). Higher scores = better verbal fluency/executive function. We report the Total Correct scaled score per the manual.
Time Frame: at baseline and 5 weeks of rTMS
Population: Subjects were randomized to receive right or left IPL stimulation.
Measure: Mean (Standard Deviation); unit: scaled score (higher = better)
Arm/Group | Left IPL Stimulation | Right IPL Stimulation
Number analyzed (Participants) | 5 | 6
scaled score (higher = better)
  Baseline | 5.8 (3.834) | 8.5 (7.778)
  Week 5 | 5.6 (2.793) | 9 (9.899)

4. Secondary Outcome: The Effects of rTMS on Executive Function Using Flanker Task
Description: NIH Toolbox Flanker Inhibitory Control and Attention; Age-Adjusted Standard Scores (mean 100, SD 15) reported. Higher scores = better inhibitory control/attention.
Time Frame: at baseline and 5 weeks of rTMS
Population: Subjects were randomized to receive right or left IPL stimulation.
Measure: Mean (Standard Deviation); unit: standard score (higher =better)
Arm/Group | Left IPL Stimulation | Right IPL Stimulation
Number analyzed (Participants) | 5 | 6
standard score (higher =better)
  Baseline | 66.8 (14.025) | 86 (22.996)
  Week 5 | 71.4 (16.742) | 83.833 (24.555)

5. Secondary Outcome: The Effects of rTMS on Executive Function
Description: NIH Toolbox Dimensional Change Card Sort (DCCS); Age-Adjusted Standard Scores (mean 100, SD 15) reported. Higher scores = better cognitive flexibility.
Time Frame: at baseline and 5 weeks of rTMS
Population: Subjects were randomized to receive right or left IPL stimulation.
Measure: Mean (Standard Deviation); unit: standard score (higher =better)
Arm/Group | Left IPL Stimulation | Right IPL Stimulation
Number analyzed (Participants) | 5 | 6
standard score (higher =better)
  Baseline | 77.4 (23.416) | 76.8 (23.784)
  Week 5 | 78.6 (17.544) | 80.2 (23.721)

ADVERSE EVENTS:
Time Frame: 3 month
Description: We had to adverse events, adverse events were monitored
Arm/Group | Left IPL Stimulation | Right IPL Stimulation
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8

LIMITATIONS AND CAVEATS:
Although we were budgeted for 20 patients, we only recruited 16 patients and 5 dropped out and did not complete behavioral measures. Fortunately, all 16 subjects completed the 10 sessions of TMS and there were no adverse effects. One of the impediments was persuading families to attend 10 sessions of TMS as well as the neuropsychic assessments.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-21): https://cdn.clinicaltrials.gov/large-docs/12/NCT05371912/Prot_SAP_000.pdf